CLINICAL TRIAL: NCT02584751
Title: Comparison of GERD and the Effects of Anti-Reflux Therapy on Pulmonary Function Between Able-Bodied and SCI Individuals
Brief Title: GERD and Anti-Reflux Therapy Between Able-bodied and SCI Individuals
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Miroslav Radulovic, M.D., Associate Researcher, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAD-16-02
Record Dates: First submitted 2015-10-09; First posted 2015-10-23 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Gastro Esophageal Reflux Disorder
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Able-Bodied non-GERD (Active Comparator): Able-bodied patients who are not diagnosed with GERD during screening will act as controls.
  Interventions: Device: 24 Hour pH Monitor; Procedure: Pulmonary Function Examination; Procedure: Exhaled Nitric Oxide; Procedure: Exhaled Breath Concentrate (EBC); Procedure: Bernstein's Acid Clearance Test; Procedure: Esophageal Motility
- SCI non-GERD (Active Comparator): SCI patients who are not diagnosed with GERD during screening will act as controls
  Interventions: Device: 24 Hour pH Monitor; Procedure: Pulmonary Function Examination; Procedure: Exhaled Nitric Oxide; Procedure: Exhaled Breath Concentrate (EBC); Procedure: Bernstein's Acid Clearance Test; Procedure: Esophageal Motility
- SCI GERD (Experimental): For those SCI subjects who are identified with GERD, they will undergo a 8week treatment of Omeprazole to reduce GERD
  Interventions: Drug: Omeprazole; Device: 24 Hour pH Monitor; Procedure: Pulmonary Function Examination; Procedure: Exhaled Nitric Oxide; Procedure: Exhaled Breath Concentrate (EBC); Procedure: Bernstein's Acid Clearance Test; Procedure: Esophageal Motility
- Able-bodied GERD (Active Comparator): For those AB subjects who are identified with GERD will act as controls. Note they will not receive treatment for GERD in this study. We will notify their primary care physician during the study so that they may receive treatment.
  Interventions: Device: 24 Hour pH Monitor; Procedure: Pulmonary Function Examination; Procedure: Exhaled Nitric Oxide; Procedure: Exhaled Breath Concentrate (EBC); Procedure: Bernstein's Acid Clearance Test; Procedure: Esophageal Motility

INTERVENTIONS:
Drug: Omeprazole — Omeprazole is a commonly prescribed anti-reflux medication. If a SCI patient has GERD, they will be prescribed with 40mg omeprazole twice daily for two months
  Arms: SCI GERD
Device: 24 Hour pH Monitor — Monitors the acidity and levels of pH in the esophagus for 24hours and helps diagnose people with GERD
Procedure: Pulmonary Function Examination — Assess pulmonary function such as lung volumes, spirometry, and max inspiration/expiration pressures.
Procedure: Exhaled Nitric Oxide — Used to measure inflammation markers for airway resistance.
Procedure: Exhaled Breath Concentrate (EBC) — EBC will be used to measure airway inflammation via specific markers, such as 8-isoprostane. This marker, if elevated, has been identified as an indicator for asthma inflammation.
Procedure: Bernstein's Acid Clearance Test — Bernstein test is a clinical test for the diagnosis of chest pain in association with gastric acid exposure
Procedure: Esophageal Motility — Esophageal Motility will be used to measure a subject's ability to swallow a bolus (i.e. saline solution) and record pressure changes throughout the esophagus during the swallow. This will also be used to identify anatomical landmarks, such as lower esophageal sphincter, which are necessary for proper placement of 24hr pH catheter.

SUMMARY:
Respiratory dysfunction, esophageal dysmotility, and a gastroesophageal reflux disease (GERD) have been demonstrated to be highly prevalent in persons with SCI. GERD has been linked to respiratory symptoms and conditions such as asthma, chronic cough, and an increased rate of respiratory infections in the general population. In persons with asthma, respiratory symptoms and dependency on asthma medications have been reduced by treatment with anti-reflux medication. Possible mechanisms have been proposed for this link, including the microaspiration of reflux materials, which may result in airway acidification and aspiration pneumonia, or the stimulation of the vagus nerve through acid-sensitive receptors in the esophagus with associated esophageal inflammation and reflex bronchoconstriction. Investigators propose to study the effects of anti-reflux therapy (proton pump inhibition) in persons with SCI on objective and subjective symptoms of respiratory function to determine the underlying mechanisms of airway inflammation due to GERD.

DETAILED DESCRIPTION:
Complete or partial loss of respiratory muscle innervation in individuals with cervical (C1-8) and high thoracic (T1-6) injuries leads to inadequate ventilation and inability to effectively clear secretions, often prompting supportive ventilation following initial injury. Development of atelectasis, pneumonias and respiratory failure are the most common respiratory complications observed during the acute phase of injury. The role of chronic airway inflammation on pulmonary function in persons with SCI is unknown, although the investigators' recent work has shown that individuals with cervical SCI have elevated levels of exhaled nitric oxide (NO), comparable to those seen in mild asthma. It is now widely believed that in the airways of asthmatic patients, the release of NO represents a physiological mechanism to counteract the bronchoconstriction caused by various stimuli. In persons with cervical SCI, bronchoconstriction may represent a consequence of unopposed parasympathetic influence, but alternative mechanisms, such as recurrent infections secondary to impaired cough effectiveness, systemic inflammatory response following SCI, or extra-esophageal manifestations of underlying esophageal dysmotility and/or GERD need to be evaluated. In general population, it has been long recognized that esophageal dysmotility and/or GERD may lead to extra-esophageal manifestations. Reflux can affect both upper and lower respiratory systems leading to the variety of extra-esophageal manifestations, such as reflux asthma, chronic cough, hoarseness, chronic sinusitis, laryngitis, loss of dental enamel, idiopathic pulmonary fibrosis, recurrent pneumonia, chronic bronchitis, etc. 2 possible mechanisms of these complications have been identified: the direct aspiration of reflux content and indirectly, stimulation of vagally-mediated reflexes. Regardless of the underlying mechanisms, treatments with acid-reducing therapies have shown improvement in GERD and extra-esophageal manifestations of the disease the general population. Investigators propose to study the effects of anti-reflux therapy (proton pump inhibition) in persons with SCI on objective and subjective symptoms of respiratory function to determine the underlying mechanisms of airway inflammation due to GERD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Tetraplegia (Level of SCI C4-8);
* Subjects with High Paraplegia (Level of SCI T1-T7);
* Subjects with Low Paraplegia (Level of SCI T8 or below);
* Able-Bodied Subjects (non SCI)
* Duration of injury ≥ 1 year; and
* Chronological age between 18-75 years.

Exclusion Criteria:

* Smoking, active or history of smoking < 6 months;
* Any history of blast injuries to the chest;
* Active respiratory disease or recent (within 3 months) respiratory infections;
* Use of medications known to alter airway caliber (i.e. beta 2 agonists or anticholinergic agents);
* Use of Protein Pump Inhibitors < 8 weeks before testing;
* Use of H2 receptor blockers <8 weeks before testing;
* History of gastrectomy;
* History of esophageal malignancy and/or resection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
DeMeester Score | 24hours
  A DeMeester score will be calculated from the 24hour pH monitoring to determine if an individual has GERD.

SECONDARY OUTCOMES:
Pulmonary Function Tests | 2days
  Pulmonary Function values and results will be compared to one another to determine if a protein pump inhibitor treatment decreases GERD and improves pulmonary function
Symptom Surveys and Questionnaires | 2days
  An 11 question survey assessing GERD and a 15 question survey assessing dysphagia or difficulty swallowing will be used to confirm diagnosis of GERD and compared across the various groups.

CONTACTS AND LOCATIONS:
Locations (1):
- James J. Peters VA Medical Center, The Bronx, New York, United States